CLINICAL TRIAL: NCT02843737
Title: Multicenter Observational Study to Validate a New Index for Sleep Fragmentation Analysis: Sleep Diversity Index (SDI)
Acronym: SDI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Toulon University (Unknown); bio N com Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: CH-2014-02 / IDS 2
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Sleep Fragmentation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Polysomnography under spontaneous breathing — Patient will come to the sleep laboratory to perform the polysomnography under spontaneous breathing prescribed by the clinician

SUMMARY:
The investigators want to validate the Sleep Diversity Index as a diagnosis tool of sleep fragmentation on 405 patients who will perform a polysomnography under spontaneous breathing.

DETAILED DESCRIPTION:
Sleep fragmentation is one of the main problems of sleep disorders especially in respiratory failure. During this last decade, several indicators of sleep fragmentation were introduced but none of them seems to take into account the succession of sleep stages. To tackle with this problem, The investigators used the Shannon entropy index for modelling sleep stages diversity from an hypnogram and for assessing more accurately sleep quality by quantifying its fragmentation. The investigators developed a new tool we called Sleep Diversity Index (SDI).

In a retrospective study, the investigators calculated Sleep diversity index for 55 healthy subjects and 56 patients with suspected sleep apnea syndrom. Using the receiver operating characteristic (ROC) curves the threshold of fragmentation was determined at 20%. If SDI is lower than 20%, then sleep is considered as non-fragmented and otherwise, sleep is considered as fragmented.

To validate our SDI it is necessary to compare this diagnosis tool to a "gold standard" based on the clinician diagnosis and a mathematical diagnosis index created from objective criteria of polysomnography. The investigators propose a multicenter study to validate the SDI as a diagnosis tool of sleep fragmentation.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous polysomnography

Exclusion Criteria:

* Insomnia
* Patients with psychoactive drug having an important effect on sleep

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who performed a spontaneous breathing polysomnography
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Comparison between mathematical analysis and clinician interpretation of polysomnographic datas recorded under spontaneous breathing | One night
  In order to determine the fragmentation of patient's sleep with two different approach and test the sleep diversity index .

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D'AMORE, MD, Principal Investigator — Centre Hospitalier Intercommunal Toulon La Seyne sur mer
Locations (3):
- France (3):
  - CHU Dijon, Dijon
  - CHU Poitiers, Poitiers
  - Centre Hospitalier Intercommunal Toulon La Seyne Sur Mer (CHITS), Toulon